CLINICAL TRIAL: NCT03085628
Title: Sex- and Context-dependent Effects of Oxytocin on Social Reward Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-08
Record Dates: First submitted 2017-03-02; First posted 2017-03-21 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Mental Health Wellness 1; Social Behavior; Emotion
Keywords: social sharing; social reward; functional magnetic resonance imaging; reward circuit
MeSH Terms: conditions — Social Behavior | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Oxytoxin nasal spray
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 40IU
  Arms: Oxytocin
Drug: Placebo — 40IU
  Arms: Placebo

SUMMARY:
The aim of the present study is to examine whether the neuropeptide oxytocin (OXT) influences social reward processing and whether the effects are context- and sex-dependent.

DETAILED DESCRIPTION:
In a double-blind, randomized, placebo-controlled, between-subject design healthy volunteers will receive either oxytocin or placebo nasal spray (40IU in 10 puffs).

Subjects will come to the experiment in pairs (two friends of the same sex). 45 min after drug administration, the two subjects will simultaneously undergo a social reward task - during the task, functional magnetic resonance imaging (fMRI) data will be acquired from one of them. During the social reward task subjects will be asked to rate the valence and arousal of emotional pictures in three different conditions: alone, share with a stranger and share with their friend.

Before treatment, subjects will complete a range of validated questionnaires to control for potential confounders, such as level of depression (assessed using the BDI) and to explore associations between relevant personality factors and treatment effects, such as adult attachment style (assessed using the AAS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorder, right-handed, had normal or corrected-to normal vision.

Exclusion Criteria:

* self-reported medication use, substance abuse, and presence of medical or psychiatric disorders

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 252 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
fMRI: neural activity during social reward processing | 45-115 minutes after administration
  Main effects of treatment will be analyzed on fMRI activity during a social reward processing paradigm.
Modulatory effects of sex on fMRI based neural indices during social reward processing | 45-115 minutes after administration
  Interaction between treatment effects and sex will be analyzed on fMRI indices acquired during reward processing
fMRI: functional connectivity during social reward processing | 45-115 minutes after administration
  Main effects of treatment will be analyzed on fMRI connectivity during a social reward processing paradigm.

SECONDARY OUTCOMES:
Behavior: arousal ratings during social reward processing | 45-115 minutes after administration
  Main effects of treatment will be analyzed on behavioral ratings of arousal acquired during the social reward processing paradigm.
Behavior: valence rating during social reward processing | 45-115 minutes after administration
  Main effects of treatment will be analyzed on behavioral ratings of valence acquired during the social reward processing paradigm.
Modulatory effects of sex on arousal ratings during social reward processing | 45-115 minutes after administration
  Interactions between treatment and sex will be analyzed on behavioral arousal ratings acquired during the social reward processing paradigm.
Modulatory effects of sex on valence ratings during social reward processing | 45-115 minutes after administration
  Interactions between treatment and sex will be analyzed on behavioral valence ratings acquired during the social reward processing paradigm.
Pre-treatment modulators: attachment style (AAS) | 45-115 minutes after administration
  Associations between neural and behavioral effects of treatment with pre-treatment attachment style as assessed by the Adult Attachment Scale (AAS)

CONTACTS AND LOCATIONS:
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma X, Zhao W, Luo R, Zhou F, Geng Y, Xu L, Gao Z, Zheng X, Becker B, Kendrick KM. Sex- and context-dependent effects of oxytocin on social sharing. Neuroimage. 2018 Dec;183:62-72. doi: 10.1016/j.neuroimage.2018.08.004. Epub 2018 Aug 4. PMID 30086408